CLINICAL TRIAL: NCT04317300
Title: The Feasibility of Treatment for Vaping Cessation
Brief Title: Feasibility of Treatment for Vaping Cessation
Acronym: VAPEscape
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: medication has not been available for the intervention
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-011437
Record Dates: First submitted 2020-02-14; First posted 2020-03-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Vaping
Keywords: electronic cigarettes; vaping; e-cigarettes
MeSH Terms: conditions — Vaping | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: 12 weeks of varenicline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E-cigarette users (Experimental): Participants who are regular users of e-cigarettes will be treated with a 12 week course of varenicline for stopping vaping.
  Interventions: Drug: Varenicline; Other: brief behavioral therapy

INTERVENTIONS:
Drug: Varenicline — Dosage of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4 to 7, and then to the maintenance dose of 1 mg twice daily for the remaining 11 weeks of treatment.
  Other Names: Chantix®
Other: brief behavioral therapy — brief behavioral therapy

SUMMARY:
Researchers are gathering information on the feasibility of treating e-cigarette users with 12-weeks of varenicline (Chantix®) in assisting with stopping the use of e-cigarettes.

DETAILED DESCRIPTION:
Because the process of developing nicotine dependence and the reinforcing mechanisms of nicotine delivered in high concentrations are similar between tobacco cigarettes and newer generation electronic cigarettes, the investigators hypothesize that evidence based treatment approaches used in treating tobacco dependence should be effective in treating dependence on electronic cigarettes. Since there is no existing evidence base for treatment of electronic cigarette dependence, preliminary evidence is needed from feasibility and open label studies to guide in the development of future randomized clinical trials. In this study, vaping participants will be treated with a 12 week course of varenicline as well as have nicotine dependence counseling through a certified tobacco treatment specialist followed up 12 weeks post end of medication.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and ≤65 years of age;
* No use of tobacco in any form (except E-cigarettes) in the past 3 months;
* currently using e-cigarettes

Exclusion Criteria:

* Current moderate or severe depression
* Use of any treatments for tobacco dependence within the past 30 days;
* Recent history (past 3 months) of abuse of, or dependence on, a substance other than nicotine;
* Women who are pregnant or lactating, or who are of childbearing potential and are likely to become pregnant during the medication phase, or a male who is able to father a child, and are not willing to use a reliable form of contraception,
* Subject describes having a medical history of: a) unstable angina; b) myocardial infarction within the past 3 months; c) coronary angioplasty; or d) an untreated cardiac dysrhythmia;
* Subject currently has cancer [excluding non-melanoma skin cancer] not in remission;
* Known allergy to varenicline;
* Subject has a medical condition deemed by the investigators to be exclusionary to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of e-cigarette abstinence after 12 weeks of treatment with varenicline plus brief behavioral therapy as an aid to stop vaping | 12 weeks
  The rate of self reported e-cigarette abstinence verified biochemically with nicotine and nicotine metabolites in urine will be assessed at the end of a 12-week course of varenicline plus brief behavioral therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Ebbert, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials